CLINICAL TRIAL: NCT02145741
Title: An Open-label Phase I Dose Escalation Trial of Weekly Intravenous Administrations of BI 836845 in Japanese Patients With Advanced Solid Tumours
Brief Title: Weekly Intravenous Administrations of BI 836845 in Japanese Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1280.15
Record Dates: First submitted 2014-05-21; First posted 2014-05-23 (Estimated); Results first posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — xentuzumab

ARMS (3):
- 750 milligram Xentuzumab (Experimental): 750 milligram Xentuzumab given weekly (days 1, 8, and 15) as an intravenous infusion over 1 hour. Patients stayed on treatment in 21-day cycles until disease progression or undue toxicities.
  Interventions: Drug: 750 milligram Xentuzumab
- 1000 milligram Xentuzumab (Experimental): 1000 milligram Xentuzumab given weekly (days 1, 8, and 15) as an intravenous infusion over 1 hour. Patients stayed on treatment in 21-day cycles until disease progression or undue toxicities.
  Interventions: Drug: 1000 milligram Xentuzumab
- 1400 milligram Xentuzumab (Experimental): 1400 milligram Xentuzumab given weekly (days 1, 8, and 15) as an intravenous infusion over 1 hour. Patients stayed on treatment in 21-day cycles until disease progression or undue toxicities.
  Interventions: Drug: 1400 milligram Xentuzumab

INTERVENTIONS:
Drug: 750 milligram Xentuzumab — 750 milligram Xentuzumab given weekly (days 1, 8, and 15) as an intravenous infusion over 1 hour. Patients stayed on treatment in 21-day cycles until disease progression or undue toxicities.
  Other Names: BI 836845
  Arms: 750 milligram Xentuzumab
Drug: 1000 milligram Xentuzumab — 1000 milligram Xentuzumab given weekly (days 1, 8, and 15) as an intravenous infusion over 1 hour. Patients stayed on treatment in 21-day cycles until disease progression or undue toxicities.
  Other Names: BI 836845
  Arms: 1000 milligram Xentuzumab
Drug: 1400 milligram Xentuzumab — 1400 milligram Xentuzumab given weekly (days 1, 8, and 15) as an intravenous infusion over 1 hour. Patients stayed on treatment in 21-day cycles until disease progression or undue toxicities.
  Other Names: BI 836845
  Arms: 1400 milligram Xentuzumab

SUMMARY:
This open-label dose escalation phase I trial, 1280.15, is with the first administration of BI 836845 in Japanese patients with various types of advanced solid tumours. The rationale behind this study is to identify the maximum tolerated dose (MTD) of BI 836845 in Japanese patients with advanced solid tumours as weekly intravenous administration.

ELIGIBILITY:
Inclusion criteria:

Patients who meet all of the following inclusion criteria by the judgment of investigator are eligible to receive the study treatment:

1. Patients with cytologically or histologically confirmed solid tumours that are refractory to standard therapy, for whom no standard therapy of proven efficacy exists, or who are not amenable to establish treatment options
2. Age >=20 years old
3. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
4. Written informed consent that is consistent with Good Clinical Practice (GCP) guidelines

Exclusion criteria:

Patients who apply any of the following exclusion criteria by the judgment of investigator are not eligible to receive the study treatment:

1. Active infectious disease to be incompatible with the study treatment
2. Patients who do not have sufficient major organ function and meet any of the following test results at screening period

   * Cardiac left ventricular function with resting ejection fraction <=50% as determined by echocardiography (ECHO) or multiple-gated acquisition scan (MUGA)
   * Absolute neutrophil count <1500/µL
   * Platelets <100 000/µL
   * Total bilirubin >1.5 × the upper limit of normal (ULN)
   * Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >2.5 × ULN (in case of known liver metastases, AST and/or ALT >5 × ULN)
   * Creatinine >1.5 × ULN
   * Haemoglobin <9 g/dL
   * HbA1c >=8% and fasting glucose >8.9 mmol/L (>160 mg/dL)
3. Serious illness or concomitant non-oncological disease including severe, acute, or chronic medical or psychiatric condition, or laboratory abnormality that may compromise the safety of the patient during the study, affect the patient's ability to complete the study, or interfere with interpretation of study results considered by the investigator to be incompatible with the study treatment
4. History of thrombosis (except tumour invading great vessels) within 1 year before start of study treatment or if concurrent anticoagulation required
5. Patients not recovered from any therapy-related toxicities from previous chemotherapies, hormonal therapies, immunotherapies, molecular-targeted therapies, or radiotherapies to Common Terminology Criteria for Adverse Events (CTCAE) grade <=1
6. Patients who have not recovered from any previous surgery and major surgery within the last 4 weeks before start of study treatment
7. Patients with untreated or symptomatic brain metastases.
8. Patients who have been treated with any of the following within 4 weeks before start of study treatment: chemotherapies, immunotherapies, radiotherapies (within 2 weeks before start of study treatment for local palliative radiotherapies for the treatment of brain metastasis or extremities), biological therapies, molecular-targeted therapies, hormonal therapies for breast cancer within 2 weeks before start of study treatment, or treatment with other investigational drugs.
9. Patients who have used any investigational drug within 4 weeks before start of study treatment or who have planned concomitantly use with the trial.
10. Patients unable to comply with the clinical trial protocol (CTP)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-06-11 (Actual); Primary Completion 2015-07-01 (Actual); Study Completion 2023-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- National Cancer Center Hospital East, Chiba, Kashiwa, Japan

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Doi T, Kuboki Y, Naito Y, Ishida M, Tanaka T, Takeuchi Y. A phase 1 trial of xentuzumab, an IGF-neutralizing antibody, in Japanese patients with advanced solid tumors. Cancer Sci. 2022 Mar;113(3):1010-1017. doi: 10.1111/cas.15231. Epub 2022 Jan 13. PMID 34870878
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an open-label study, with a dose escalation cohort according to a 3+3 design followed by an expansion cohort.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- 750 Milligram Xentuzumab (BI 836845): 750 milligram Xentuzumab (BI 836845) given weekly (days 1, 8, and 15) as an intravenous infusion over 1 hour. Patients stayed on treatment in 21-day cycles until disease progression or undue toxicities.
- 1000 Milligram Xentuzumab (BI 836845): 1000 milligram Xentuzumab (BI 836845) given weekly (days 1, 8, and 15) as an intravenous infusion over 1 hour. Patients stayed on treatment in 21-day cycles until disease progression or undue toxicities.
- 1400 Milligram Xentuzumab (BI 836845): 1400 milligram Xentuzumab (BI 836845) given weekly (days 1, 8, and 15) as an intravenous infusion over 1 hour. Patients stayed on treatment in 21-day cycles until disease progression or undue toxicities.
Period: Overall Study
Arm/Group | 750 Milligram Xentuzumab (BI 836845) | 1000 Milligram Xentuzumab (BI 836845) | 1400 Milligram Xentuzumab (BI 836845)
Started | 6 | 9 | 6
Maximum Tolerated Dose (MTD) Set | 3 | 3 | 6
Completed | 0 | 3 | 0
Not Completed | 6 | 6 | 6
Not completed — Progressive disease | 3 | 6 | 6
Not completed — quality issue with the administered drug | 3 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set - This patient set included all patients who were documented to have received and taken at least 1 dose of trial medication during the treatment cycles since Day 1.
Groups:
- Total: Total of all reporting groups
Arm/Group | 750 Milligram Xentuzumab (BI 836845) | 1000 Milligram Xentuzumab (BI 836845) | 1400 Milligram Xentuzumab (BI 836845) | Total
Number analyzed (Participants) | 6 | 9 | 6 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.33 (10.82) | 52.00 (16.58) | 64.67 (9.16) | 58.00 (21.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 1 | 8
  Male | 2 | 6 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 9 | 6 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 6 | 9 | 6 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Xentuzumab in Japanese Patients With Advanced Solid Tumours, as Identified by the Number of Patients With Dose-limiting Toxicities (DLTs)
Description: MTD of xentuzumab in Japanese patients with advanced solid tumours, as identified by the number of patients with DLTs. The MTD of xentuzumab was defined as the highest dose tested with DLT occurring in not more than 1 out of 6 evaluable patients.
  DLTs were defined as:
  Haematological toxicities:
  Common Terminology Criteria for Adverse Events (CTCAE) grade (g) 4 neutropenia ≥7 days (d), select cases of Febrile neutropenia, Infections or CTCAE g4 thrombocytopenia or CTCAE g3 thrombocytopenia.
  Non-haematological toxicities:
  CTCAE grade 3 or 4 non-haematologic toxicity, with exceptions CTCAE grade≥2 infusion reaction or nausea and/or vomiting with exceptions CTCAE grade ≥3 skin toxicity, hyperglycaemia, any electrolyte adverse events (AE), fatigue or asthenia with exceptions No recovery from a non-DLT CTCAE g≥3 toxicity to g≤1 within 14 d of administered dose Other drug-related AEs (CTCAE g2), might qualify as a DLT, which will be determined on a case by case bases.
Time Frame: During the first cycle of treatment, up to 21 days of treatment.
Population: The Maximum tolerated dose (MTD) set was defined as the set of patients that were fully evaluable for the MTD in the first treatment cycle.
Measure: Number; unit: Milligram
Groups:
- Xentuzumab (BI 836845): Comprises all dose cohorts (750, 1000 and 1400 milligram) in the dose escalation cohort. Xentuzumab (BI 836845) given weekly (days 1, 8, and 15) as an intravenous infusion over 1 hour. Patients stayed on treatment in 21-day cycles until disease progression or undue toxicities.
Arm/Group | Xentuzumab (BI 836845)
Number analyzed (Participants) | 12
Milligram | NA — There were no dose-limiting toxicities experienced by any patient during the MTD evaluation period, thus MTD was not reached.

ADVERSE EVENTS:
Time Frame: Adverse events collection: From first day of treatment until the last day of treatment + the residual effect period (42 days), up to 1499 days. All-cause mortality: From start of study till the end of study, up to 1527 days.
Description: Treated set - This patient set included all patients who were documented to have received and taken at least 1 dose of trial medication during the treatment cycles since Day 1.
Arm/Group | 750 Milligram Xentuzumab (BI 836845) | 1000 Milligram Xentuzumab (BI 836845) | 1400 Milligram Xentuzumab (BI 836845)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/9 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 3/9 | 0/6
Other Adverse Events (participants affected / at risk) | 3/6 | 9/9 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 750 Milligram Xentuzumab (BI 836845) (N=6) | 1000 Milligram Xentuzumab (BI 836845) (N=9) | 1400 Milligram Xentuzumab (BI 836845) (N=6)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 750 Milligram Xentuzumab (BI 836845) (N=6) | 1000 Milligram Xentuzumab (BI 836845) (N=9) | 1400 Milligram Xentuzumab (BI 836845) (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 4 | 1
Nausea (Gastrointestinal disorders) | 0 | 4 | 1
Fatigue (General disorders) | 1 | 4 | 1
General physical health deterioration (General disorders) | 0 | 0 | 1
Malaise (General disorders) | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 3 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 0
C-reactive protein increased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1 | 0
White blood cell count decreased (Investigations) | 1 | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Eustachian tube patulous (Ear and labyrinth disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Corneal disorder (Eye disorders) | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 0
Ocular hypertension (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 2 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 0
Toothache (Gastrointestinal disorders) | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0
Influenza like illness (General disorders) | 0 | 3 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 2 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 0
Helicobacter infection (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Fractured coccyx (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Monoparesis (Nervous system disorders) | 0 | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-04-29): https://cdn.clinicaltrials.gov/large-docs/41/NCT02145741/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT02145741/SAP_001.pdf